CLINICAL TRIAL: NCT02082249
Title: An Open-Label Three-Part Extension Study Assessing Safety, Tolerability and Efficacy of ABT-SLV187 in Subjects With Advanced Parkinson's Disease and Persistent Motor-Complications Despite Optimized Treatment With Available Anti-Parkinsonian Medications
Brief Title: An Extension Study to Assess the Safety, Tolerability and Efficacy of ABT-SLV187 in Subjects With Advanced Parkinson's Disease and Persistent Motor-Complications Despite Optimized Treatment With Available Anti-Parkinsonian Medications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-923
Record Dates: First submitted 2014-02-14; First posted 2014-03-10 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Advanced Parkinson's Disease
Keywords: Safety; Tolerability; Efficacy; levodopa-carbidopa intestinal gel; levodopa; carbidopa; Advanced Parkinson's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABT-SLV187 (Experimental): up to 6 years
  Interventions: Drug: ABT-SLV187

INTERVENTIONS:
Drug: ABT-SLV187 — Dose levels will be individually optimized

SUMMARY:
This is an extension study to evaluate the long-term safety and tolerability of ABT-SLV187 in subjects with advanced Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects completing 12 weeks treatment in Study M12-921 who would benefit from long-term treatment from ABT-SLV187. Alternatively, subjects who (i) participated in the Phase 2 Study M12-925 (ii) would, in the opinion of the Investigator, benefit from ABT-SLV187 treatment in the Study M12-923, (iii) did not discontinue the M12-925 Study due to safety reason, and (iv) meet all entry requirements. Lastly, subjects who completed another ABT-SLV187 study (e.g., Study M12-927) in South Korea.
2. The subject must be able to understand the nature of the study and must provide written informed consent prior to the conduct of any study procedures (including any changes occurring in the subject's current therapeutic regimen).
3. The subject must be willing to continue on treatment.

Exclusion Criteria:

1. Subject is enrolled in another clinical trial.
2. Psychiatric, neurological or behavioral disorders that may interfere with the ability of subjects to give informed consent, or interfere with the conduct of the study.
3. Medical, laboratory, or surgical issues deemed by the Investigator to be clinically significant and in the opinion of the PI, would be a contraindication to continued levodopa therapy.
4. Uncooperative attitude or reasonable likelihood for non-compliance with the protocol.
5. Subject has current significant suicidal ideation as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale completed at the Week 12 Visit of Study M12-921 or at the Baseline Visit of the current study for M12-925 or M12-927 study subjects.
6. Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to continue to receive ABT-SLV187.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | From Day 1 up to 6 years (estimated maximum)
  All negative changes in health during the study will be treated and recorded during the study.

SECONDARY OUTCOMES:
Change in Patient Global Impression of Change (PGIC) scores | From Screening Visit 2 of M12-921 to Week 52 of M12-923
  The PGIC is a 7-point response scale. The subject will be asked by the Investigator or qualified designee to rate their change in their disease status.
Change in the Unified Parkinson's Disease Rating Scale (UPDRS) score | From Day 1 up to 36 months (estimated maximum)
  The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the course of Parkinson's disease.
Change in the Parkinson's Disease Questionnaire-39 (PDQ-39) scores | From Screening Visit 2 of M12-921 to Week 52
  The PDQ-39 is a disease-specific instrument designed to measure aspects of health that are relevant to subjects with PD, and which may not be included in general health status questionnaires.
Change in PD Diary mean daily "On" time without troublesome dyskinesia ("On" time without dyskinesia or with non-troublesome dyskinesia) or "On" time with troublesome dyskinesia | From Day 1 to Week 52
  The study will assess the difference in the amount of time a subject is able to move and function well during the day.
Change in the mean daily "Off" time (hours) as measured by the Parkinson's Disease (PD) Diary © | From Day 1 to Week 52
  The study will assess the difference in the amount of time a subject is unable to move and function during the day.
Change in Clinical Global Impression of Change (CGI-C) scores | From Screening Visit 2 of M12-921 to Week 52 of M12-923
  The 7-item CGI-C (Change) scale assesses the overall degree of illness relative to Week 0. A rating of 4 is equivalent to "no change." Ratings < 4 are equivalent to "improvement" and ratings of 4 are equivalent to "worsening."

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (7):
- Japan (5):
  - National Hospital Organization Asahikawa Medical Center /ID# 101178, Asahikawa, Hokkaido
  - National Hospital Organization Sagamihara National Hospital /ID# 98662, Sagamihara-shi, Kanagawa
  - Osaka University Hospital /ID# 108335, Suita-shi, Osaka
  - National Center of Neurology and Psychiatry /ID# 98664, Kodaira, Tokyo
  - Kyoto University Hospital /ID# 112136, Sakyo-ku
- Seoul National University Hospital /ID# 105935, Seoul, South Korea
- Linkou Chang Gung Memorial Ho /ID# 102297, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Murata M, Mihara M, Hasegawa K, Jeon B, Tsai CH, Nishikawa N, Oeda T, Yokoyama M, Robieson WZ, Chatamra K, Facheris MF, Benesh J. Safety and efficacy of levodopa-carbidopa intestinal gel: results from an open-label extension study in Japanese, Korean and Taiwanese patients with advanced Parkinson's disease. Ther Adv Neurol Disord. 2018 Feb 26;11:1756286418759315. doi: 10.1177/1756286418759315. eCollection 2018. PMID 29511383
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/levodopa_carbidopa_M12-923.pdf